CLINICAL TRIAL: NCT04399278
Title: End-eXpiratory Occlusion Test to Predict fluId REsponsiveness in the Operating Room: Prospective Randomized Clinical Trial Comparing Two Occlusion Tests (EXPIRE)
Brief Title: End-eXpiratory Occlusion Test to Predict fluId REsponsiveness in the Operating Room (EXPIRE)
Acronym: EXPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EXPIRE - RBHP 2020 FUTIER
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hemodynamic Instability; General Anesthesia; Surgery; Protective Mechanical Ventilation
Keywords: End-expiratory occlusion; Fluid responsiveness; Fluid Challenge; Intraoperative monitoring; Hemodynamic optimization

STUDY DESIGN:
Intervention Model Description: The EEO test will be performed by interrupting the mechanical ventilation at end-expiration over 15 and 30 seconds using the end-expiratory hold button available on the anesthesia ventilator. Each occlusion will be separated by 1 minute to allow a return to the baseline value.
  Hemodynamic variables will be recorded before and immediately after each EEO procedure, and after a fluid challenge (4 ml/kg of 0.9% saline over 5 minutes).
  Fluid responders will be defined by an increase in stroke volume ≥15% 1 min after the end of the fluid challenge.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomization sequence by permuted blocks (random block sizes) with an allocation of 1:1 will be generated by a computer program (Stata software, version 15, StataCorp, College Station, US) The group assignment will be concealed until arrival in the operating room so that only the anesthesiologist in charge of the patient will aware to the randomization group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): The EEO test will be applied first over 15 seconds and secondly over 30 seconds (each EEO test separated by 1 minute wash-out period)
  Interventions: Diagnostic Test: Diagnostic Test: end-expiratory occlusion (EEO) test
- Group B (Other): The EEO test will be applied first over 30 seconds and secondly over 15 seconds (each EEO test separated by 1 minute wash-out period)
  Interventions: Diagnostic Test: Diagnostic Test: end-expiratory occlusion (EEO) test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: end-expiratory occlusion (EEO) test — A set of respiratory and hemodynamic measurements (including cardiac output) will be recorded at each stage:
  * T0: baseline.
  * T1: At the end of the first EEO (15 sec or 30 sec)
  * T2: 1 minute after completion of the first EEO. Return to baseline.
  * T3: At the end of the second EEO (15 sec or 30 sec)
  * T4: 1 minute after completion of the second EEO. Return to baseline.
  * T5: Before the fluid challenge test (4 ml/kg of 0.9% saline over 5 min)
  * T6: 1 minute after the end of the fluid challenge
  A first set of measurements will be performed after intubation (before the surgical incision) and will be repeated, if necessary, in case of further decrease in stroke volume during surgery or in case of any clinical indication of volume expansion (i.e., arterial persistent hypotension, major hemorrhage, etc.).

SUMMARY:
The purpose of the study is to evaluate the influence of different durations of the end-expiratory occlusion test to predict fluid responsiveness in mechanically ventilated patients in the operating room.

DETAILED DESCRIPTION:
The reduction of postoperative complications is an essential aspect of care in perioperative medicine.

Many studies have shown that individualized hemodynamic therapy, by optimizing fluid administration and cardiac output, can reduce the risk of postoperative morbidity and mortality.

A fluid challenge, consisting in the administration of a small bolus of intravenous volume of fluid over a short period of time, is one of the commonest therapeutic hemodynamic intervention to test the preload reserve and the cardiac response to an increase in intravascular volume of a patient (fluid responsiveness). However, an increase in stroke volume (or cardiac output) is only achieved in 30 to 50% of patients after a fluid challenge test. Several dynamic tests have been described to predict the response to fluid challenge, however their limits are numerous.

The end-expiratory occlusion (EEO) test, consisting in a brief interruption of mechanical ventilation at end-expiration, by preventing the variation in intra-thoracic pressure, allows an increase in venous return, cardiac preload and stroke volume. Thus, an increase in stroke volume during an EEO can predict fluid responsiveness, simulating a fluid challenge though avoiding the administration of possibly unnecessary fluids.

The EEO test has already been successfully evaluated in several studies in ICU patients. Only few studies were conducted in the operating room, with conflicting findings: one study, consisting of an EEO test of 30 seconds found that changes in stroke volume during an EEO can predict fluid responsiveness, whereas another one, consisting of an EEO test of 15 seconds did not.

The purpose of the study is to evaluate the influence of the duration of EEO test to predict fluid responsiveness in mechanically ventilated patients in operating room.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >18 years)
* Scheduled to undergo planned surgery under general anesthesia
* Surgery requiring invasive arterial and stroke volume monitoring
* Clinical indication to perform a fluid challenge
* Patients able to give informed consent
* Affiliated to a social security scheme

Exclusion Criteria:

* Patient refusal to participate or inability to provide informed consent
* Protected major
* History of lobectomy or pneumectomy
* Patient with reduced left (ejection fraction < 45%) or right ventricular systolic function
* Arrythmia
* Severe valvulopathy
* Body Mass Index <15 or > 40kg/m2
* Contraindication to insertion of invasive arterial line into radial artery
* Emergency surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
To compare the ability of an EEO over 30 sec with that of an EEO over 15 sec to predict fluid responsiveness | During surgery
  Comparison of the areas under the ROC (Receiver Operating Characteristic) curves.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Futier, PhD, Study Chair — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France